CLINICAL TRIAL: NCT05839392
Title: Novel Approaches to Target MECOM/EVI1 in Acute Myeloid Leukemia
Brief Title: Novel Approaches to Target MECOM/EVI1 in AML
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AML2623
Record Dates: First submitted 2023-04-21; First posted 2023-05-03 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: AML, Adult
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — MDS1 and EVI1 Complex Locus Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Biological characterization of AML with MECOM or atypical 3q26 rearrangements — Peripheral blood and bone marrow withdrawal

SUMMARY:
This is an academic, no-profit, multicenter, biological, non-pharmacologic study aimed at characterizing genome, transcriptome and proteome of patients affected by AML with MECOM or atypical 3q26 rearrangements.

DETAILED DESCRIPTION:
This is an academic, no-profit, multicenter, biological, non-pharmacologic study aimed at characterizing genome, transcriptome and proteome of patients affected by AML with MECOM or atypical 3q26 rearrangements. To this end, BM samples and formalin fixed/paraffin-embedded BM biopsies will be collected at enrolment, before and after treatment, at relapse.

ELIGIBILITY:
Inclusion Criteria:

* AML with MECOM or atypical 3q26 rearrangements.
* Age ≥18.
* Signed written informed consent according to ICH/EU/GCP and national local laws.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-12-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Identification of MECOM/EVI1 regulators or downstream effectors potentially druggable | At baseline
  To assess the number of regulators or effectors of MECOM/EVI1

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Roti, Principal Investigator — Department of Medicine and Surgery, University of Parma, Parma
Locations (1):
- Ematologia, Piacenza, Italy

IPD SHARING:
Plan to Share IPD: No